CLINICAL TRIAL: NCT06256224
Title: Toripalimab Combined With Definitive Chemoradiotherapy for Locally Advanced Cervical Squamous Cell Carcinoma Patients
Brief Title: Toripalimab Combined With Definitive CCRT for LACC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Haoping Xu, Prof, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024（022）
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; Chemoradiotherapy; Immunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab+CCRT (Experimental): External beam radiotherapy (EBRT) of 45-50.4Gy was delivered using intensity modulated radiation therapy (IMRT) technique to the pelvic ± para-aortic fields in 25-28 fractions, 5 days a week and was followed by brachytherapy of 24-30Gy in 3-5 fractions, once a week. Concurrent chemotherapy of cisplatin, with a dose of 40 mg/m2 by intravenous infusion, was administered once a week for 5 weeks during EBRT.
  Toripalimab 240mg by intravenous infusion was administered every 3 weeks for 6 months and maintained upto 2 years for those whose lesions did not reach complete remission at six-month follow-up.
  Interventions: Drug: Toripalimab; Radiation: CCRT
- CCRT (Active Comparator): EBRT of 45-50.4Gy was delivered using IMRT technique to the pelvic ± para-aortic fields in 25-28 fractions, 5 days a week and was followed by brachytherapy of 24-30Gy in 3-5 fractions, once a week. Concurrent chemotherapy of cisplatin, with a dose of 40 mg/m2 by intravenous infusion, was administered once a week for 5 weeks during EBRT.
  Interventions: Radiation: CCRT

INTERVENTIONS:
Drug: Toripalimab — Toripalimab combined with CCRT
  Arms: Toripalimab+CCRT
Radiation: CCRT — CCRT includes cisplatin (40 mg/m2, once a week for 5 weeks), radiotherapy (45-50.4Gy/25-28Fx, 5 fractions a week, followed by brachytherapy 24-30Gy/3-5Fx)

SUMMARY:
Cervical cancer constitutes a significant health burden for women globally. While most patients with early-stage disease can be cured with radical surgery or chemoradiotherapy, patients with high-risk locally advanced disease or with recurrent/metastatic disease have a poor prognosis with standard treatments. Immunotherapies are a rational treatment for this HPV-driven cancer that commonly expresses programmed cell death ligand-1. Toripalimab, a humanized immunoglobulin G4 monoclonal antibody against PD-1, showed promising anti-tumor efficacy in multiple solid tumors. This randomised study is evaluating toripalimab combined with CCRT versus CCRT alone for treatment-naïve LACC.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old females
* had newly diagnosed and previously untreated locally advanced squamous cell carcinoma of the uterine cervix
* FIGO 2018 stage IB3 to IVA with no evidence of distant metastasis
* ECOG PS 0-1 without major organ failure
* signed informed consent voluntarily

Exclusion Criteria:

* previously suffered from immunodeficiency disorders
* had any condition that researchers believed to be associated with increased risk of treatment
* Previously received or currently receiving other PD-1 antibody treatments or other immunotherapies targeting PD-1/PD-L1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | 2 year
  the date of the treatment to the date of disease progression or death from any cause in the absence of progression

SECONDARY OUTCOMES:
2-year local control | 2 year
  absence of disease in the cervix (uterus), upper vagina or parametria on clinical examination, imaging, and biopsy
2-year local regional control | 2 year
  absence of disease in the cervix (uterus), upper vagina or parametria and regional lymph nodes on clinical examination, imaging, and biopsy
2-year overall survival | 2 year
  the time from the start of treatment until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Haoping Xu, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No